CLINICAL TRIAL: NCT05035459
Title: Impact of B-lines-guided Intensive Heart Failure Management on Outcome of Discharged Heart Failure Patients With Residual B-lines
Brief Title: B-lines-guided Heart Failure Management in Heart Failure Patients
Acronym: IMP-OUTCOME
Status: Active, not recruiting | Type: Observational
Sponsor: Xiangtan Central Hospital (Other)
Responsible Party: Principal Investigator, Jianping Zeng, Dean, Xiangtan Central Hospital ,Director of cardiovascular clinic, Clinical Professor, Xiangtan Central Hospital
Other Study IDs: XiangtanCH
Record Dates: First submitted 2021-08-25; First posted 2021-09-05 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Lung Ultrasound; Heart Failure
Keywords: subclinical heart failure; B-line; pulmonary congestion; outcome
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Conventional heart failure management group: Patients with ≥ 3 B-lines will be divided into the conventional heart failure management group and the LUS-BL-guided intensive heart failure management group at 1:1 ratio. Patients in the conventional heart failure management group will receive conventional guideline recommended HF therapy post discharge and be followed up at 2-month interval post discharge by clinical visit. LUS-BL will be assessed at 2-month interval post discharge also in this group, but results will be enveloped.
  Interventions: Diagnostic Test: lung ultrasound
- LU-BL guided intensive heart failure management group: The group with ≥ 3 B-lines will be divided into the conventional heart failure management group and the LUS-BL-guided intensive heart failure management group at 1:1 ratio. Patients in the LUS-BL-guided intensive heart failure management group will receive optimized HF medication and medication will be adjusted according the status of LUS-BL during the follow-up at 2-month interval.
  Interventions: Diagnostic Test: lung ultrasound

INTERVENTIONS:
Diagnostic Test: lung ultrasound — drug adjustment based on lung ultrasound results
  Other Names: intensive HF management
Diagnostic Test: Lung ultrasound — drug adjustment independent on lung ultrasound results
  Other Names: conventional HF management

SUMMARY:
Background：About 50% of subclinical heart failure (Sub-HF) patients might have residual lung ultrasound B-lines (LUS-BL). Sub-HF is insensitive to widely used imaging examinations, like x-ray or echocardiography, but lung ultrasound (LUS) can sufficiently detect pulmonary congestion in Sub-HF patients. Previous studies showed that residual LUS-BL is associated worse clinical outcome among patients with chronic heart failure. In this trial, we sought to evaluate the impact of LUS-BL guided intensive HF management post discharge in patients with residual LUS-BL on outcome up to 1 year after discharge.

Aim: IMP-OUTCOME is a prospective, single-center, observational cohort study, which is designed to investigate whether LUS-BL-guided intensive HF management post discharge might improve the outcome of HF patients with residual B-lines at discharge up to 1 year after discharge.

Methods and results: After receiving the standardized treatment of HF according to current guidelines, 320 HF patients with ≥ 3 B-lines (LUS-BL, assessed within 48 hours before discharge) will be divided into the conventional HF management group and the LUS-BL-guided intensive HF management group at 1:1 ratio. LUS-BL-guided intensive HF management group will receive optimized HF medication according to current guidelines and medication will be adjusted according the status of LUS-BL in addition to symptom and physical examination results during the follow-up at 2-month interval. Patient-related clinical data including sex, age, blood chemistry, imaging examination, drug utilization, and so on will be obtained and analyzed. Following discharge from the hospital, patients in the conventional HF management group will receive optimized HF medication according to current guidelines and medication will be adjusted without knowing the status of LU-BL during the follow-up at 2-month interval. LUS-BL will be assessed at 2-month interval post discharge in both groups, results will be transferred to HF nurses, who will decide to present the LUS-BL results to managing cardiologist or envelope the LUS-BL results till study end according to group assignment. Echocardiography examination will be performed at 12 months for all patients and EF, E/e', LA size and systolic pulmonary artery pressure will be assessed. The primary endpoint is the composite of re-hospitalization for worsening HF and all-cause death during follow-up. Secondary endpoints include the change in the Duke Activity Status Index (DASI) and NT-pro BNP, arrythmia and 6-minutes walk distance at each follow up, EF and B-lines changes at final follow up. Safety profile will be noted and analyzed. Primary results will be available by early 2024.

Conclusion: This trial will clarify the impact of LUS-BL guided intensive HF management on outcome for discharged patients with residual B-lines up to 1 year after discharge in the era of sodium-glucose cotransporter-2 inhibitors and angiotensin receptor blocker-neprilysin inhibitor.

ELIGIBILITY:
Inclusion Criteria:

Hospitalized heart failure patients with objective heart failure evidence during or before hospitalization.

New York Heart Association (NYHA) class II, III, or IV.

Patients with NT-proBNP level of at least 600pg/meal (or ≥400 pg/meal if they had been hospitalized for heart failure within the previous 12 months). Atrial fibrillation or atrial flutter patients with NT-proBNP level of at least 900 pg/ml, regardless of their history of HF hospitalization.

Exclusion Criteria:

Exclusion criteria included patients with life expectancy less than 1 year due to malignancy. Patients with ARDS and pneumonia. Patients with interstitial lung disease/pulmonary fibrosis and patients on dialysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient volunteered for the trial.
Sampling Method: Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2022-03-25 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2024-08-25 (Estimated)

PRIMARY OUTCOMES:
The primary outcome consisted of readmission for worsening heart failure, or death during follow-up. | The patients will be followed up for 1 year after they were discharged from the hospital.
  follow-up by clinical visit

SECONDARY OUTCOMES:
Change the Duke Activity Status Index (DASI) score | Baseline, 2, 4, 6, 8, 10 and 12 months post discharge
  The scale consists of 12 items covering major daily physical activities such as living, housework, walking, sexual function, and recreation, and patients are judged to be able to complete the activity content by themselves. Each entry has a different score based on the weight it takes to expend on exercise energy, with the scale summing from 0 to 58.2, with higher scores representing better physical activity status.
Change in NT-proBNP | Baseline, 2, 4, 6, 8, 10 and 12 months post discharge
  pg/ml
Change in 6-minute walk distance values (6MWD) | Baseline, 2, 4, 6, 8, 10 and 12 months post discharge
  walk distance (meter)
Change in arrythmia | Baseline, 2, 4, 6, 8, 10 and 12 months post discharge
  ECG results will be evaluated and arrythmia will be evaluated

OTHER OUTCOMES:
Safety outcome | Baseline, 2, 4, 6, 8, 10 and 12 months post discharge
  * number of hospitalisation for hypotension
  * number of hospitalisation for worsening of renal function
  * number of hyperkalaemia
  * number of hypokalaemia
  * number of worsening of renal function
  * number of ketoacidosis
  * number of drug allergy
  * number of lower limb edema
  * number of severe liver dysfunction
  * number of hypoglycemia

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangtan Central Hospital, Xiangtan, Hunan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Platz E, Lewis EF, Uno H, Peck J, Pivetta E, Merz AA, Hempel D, Wilson C, Frasure SE, Jhund PS, Cheng S, Solomon SD. Detection and prognostic value of pulmonary congestion by lung ultrasound in ambulatory heart failure patients. Eur Heart J. 2016 Apr 14;37(15):1244-51. doi: 10.1093/eurheartj/ehv745. Epub 2016 Jan 26. PMID 26819225
- [Derived] Zhu Y, Li N, Wu M, Peng Z, Huang H, Zhao W, Yi L, Liao M, Liu Z, Peng Y, Zhou Y, Lu J, Li G, Zeng J. Impact of B-lines-guided intensive heart failure management on outcome of discharged heart failure patients with residual B-lines. ESC Heart Fail. 2022 Aug;9(4):2713-2718. doi: 10.1002/ehf2.13988. Epub 2022 May 20. PMID 35595501